CLINICAL TRIAL: NCT01690234
Title: Early Coordinated Multidisciplinary Intervention to Prevent Sickness Absence and Labor Market Exclusion in Patients With Low Back Pain. A Randomized Controlled Trial
Brief Title: Early Coordinated Multidisciplinary Intervention to Prevent Sickness Absence and Labor Market Exclusion in Patients With Low Back Pain.
Acronym: TIKI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Back and Rehabilitation Center, Copenhagen (Other Government)
Responsible Party: Principal Investigator, Tom Petersen, Physiotherapist, Back and Rehabilitation Center, Copenhagen
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: H-C-2008-112
Record Dates: First submitted 2012-09-19; First posted 2012-09-21 (Estimated); Last update posted 2012-09-21 (Estimated); Status verified 2012-09

CONDITIONS: Low Back Pain
Keywords: Low back pain; Return to work; Sickness absence; Rehabilitation; Multidisciplinary intervention
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Multidisciplinary intervention (Experimental): Early coordinated multidisciplinary intervention. Physiotherapist, chiropractor, rheumatologist, psychologist, occupational physician, ergonomist and social worker/case manager.
  Interventions: Procedure: Multidisciplinary intervention
- Usual care (Active Comparator): Intervention from physiotherapist, chiropractor, rheumatologist and social worker.
  Interventions: Procedure: Usual care

INTERVENTIONS:
Procedure: Multidisciplinary intervention — Early coordinated multidisciplinary intervention. Physiotherapist, chiropractor, rheumatologist, psychologist, occupational physician, ergonomist and social worker/case manager.
  Arms: Multidisciplinary intervention
Procedure: Usual care — Intervention from physiotherapist, chiropractor, rheumatologist and social worker.
  Arms: Usual care

SUMMARY:
In Denmark the number of patients, sick listed for more than four weeks is increasing, and patients suffering from musculoskeletal disorders make one third of the total amount of long-term absenteeism. Compared to other diagnoses, patients suffering from musculoskeletal diseases, including low back pain, are less likely to return to work after a period of sick leave. It seems that a multidisciplinary intervention, including cooperation between the health sector, the social sector and in the work place, has a positive effect on days off work due to musculoskeletal disorders and particularly low back pain. The aim of this study is to evaluate the effect of a work oriented multidisciplinary intervention.

A randomized controlled trial will include 770 patients with low back pain. The study population consists of patients, who are sick listed or at risk of sick leave due to LBP.

The control group is treated with usual care in a team with participation of a physiotherapist, a chiropractor, a rheumatologist and a local employed social worker The Intervention group is treated with usual care and in addition intervention of a psychologist, an occupational physician, an ergonomist and a social worker from the local sickness benefit office. The treating physiotherapist will be the RTW-coordinator. Outcome will be reported at the end of treatment as well as 6 and 12 months follow up. The primary outcome is number of days of work. Secondary outcomes are disability, pain, and quality of life.

This large RCT study is testing the effectiveness of a preventive intervention targeting patients on short term sick leave or at risk being sick listed because of low back pain. We have developed a novel multidisciplinary team structure using the treating physiotherapist as the return to work coordinator, and having the case manager from the sickness benefit office participating in team meetings.

ELIGIBILITY:
Inclusion Criteria:

* Working age adults 18-65
* Low back pain (longer than 2 weeks)
* Sicklisted or at risk
* Employed or unemployed

Exclusion Criteria:

* Severe comorbidity
* Pregnancy
* Difficulties in reading Danish language
* Application for early retirement

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 770 (Estimated)
Dates: Start 2009-09; Primary Completion 2012-09 (Actual); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Number of days off work | 12 months

SECONDARY OUTCOMES:
Disability | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Tom Petersen, PT, PhD, Principal Investigator — Back and Rehabilitaion Center Copenhagen; Annette Fisker, PT, PhDstud, Principal Investigator — University of Copenhagen, Department of Public Health
Locations (1):
- Back and Rehabilitation Center Copenhagen, Copenhagen, Copenhagen, Denmark

REFERENCES:
- [Derived] Fisker A, Langberg H, Petersen T, Mortensen OS. Effects of an early multidisciplinary intervention on sickness absence in patients with persistent low back pain-a randomized controlled trial. BMC Musculoskelet Disord. 2022 Sep 10;23(1):854. doi: 10.1186/s12891-022-05807-7. PMID 36088313
- [Derived] Fisker A, Langberg H, Petersen T, Mortensen OS. Early coordinated multidisciplinary intervention to prevent sickness absence and labour market exclusion in patients with low back pain: study protocol of a randomized controlled trial. BMC Musculoskelet Disord. 2013 Mar 13;14:93. doi: 10.1186/1471-2474-14-93. PMID 23496897